CLINICAL TRIAL: NCT00375570
Title: An Open Label, Multi-Centre, Phase III, Subject Initiated Safety Study of ME-609 in Treatment of Recurrent Herpes Simplex Labialis in Adolescents
Brief Title: Safety Study of ME-609 for Treatment of Herpes Simplex Labialis in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Borje Darpo, MD, PhD, Medivir AB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 609-07
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis | interventions — ME 609

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ME-609
  Interventions: Drug: ME-609

INTERVENTIONS:
Drug: ME-609 — Topical treatment 5 times daily for 5 days

SUMMARY:
The Purpose of this study is to evaluate the safety of ME-609 for the treatment of recurrent herpes labialis in adolescents.

DETAILED DESCRIPTION:
The objective of the study was to evaluate the safety of ME-609 for the treatment of herpes labialis recurrences in immunocompetent adolescents, 12 - 17 years of age, following a 5-day treatment with 5-time daily topical administration.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* History of recurrent herpes labialis with at two recurrences during the last twelve months

Exclusion Criteria:

* Treatment with systemic or topical antiviral agents or steroids within two weeks prior to inclusion
* Significant skin condition that occur in the area of herpes recurrences
* Nursing or/and pregnancy
* Immunosupressed state due to underlying disease (e.g. HIV infection or concomitant treatment (e.g. cancer chemotherapy)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 254 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 3 weeks after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Anders Strand, MD PhD, Principal Investigator — Department of Medical Sciences, Dermatology and Venereology University Hospital, Uppsala, Sweden